CLINICAL TRIAL: NCT04391426
Title: Analysis of Biliary Microbiota in Hepatobiliopancreatic Diseases Compared to Healthy People [MICROBILIO]
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alberto Meyer, MD PhD FACS, Principal Investigator, University of Sao Paulo
Other Study IDs: 29547920.9.0000.0068
Record Dates: First submitted 2020-04-25; First posted 2020-05-18 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Diseases; Microbiota; Early Detection of Cancer; Dysbiosis; Biliary Tract Diseases
MeSH Terms: conditions — Pancreatic Diseases; Dysbiosis; Biliary Tract Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who will undergo ERCP (case group)
- Living liver transplantation donors (control group)

SUMMARY:
The performance of the microbiota is observed in all clinical and pathological stages of carcinogenesis, since its development, diagnosis and treatment, including prognosis and survival. However, it was found that there is a scarcity of studies on biliary microbiota and its relationship with hepatobiliopancreatic diseases. Therefore, further investigation is necessary, since reaching the biliary microbiota may suggest ways for studies of biomarkers, diagnoses, tests and therapies in hepatobiliopancreatic diseases. For this, bile samples will be collected in cases and controls patients to characterize the microbiota and its variations according to the disease.

ELIGIBILITY:
Inclusion Criteria:

Endoscopic retrograde cholangiopancreatography (ERCP) candidates (case group)

* Patients over 18 years old complete
* Patients previously scheduled for ERCP
* Cannulation of the bile duct, via the transpapillary route, with the aid of a papillotome with an end kept sterile until contact with the papilla

Liver transplant living-donor (control group)

* Patients over 18 years old up to 55 years
* Previously selected patients with scheduled surgery
* BMI: 18 kg / m² to 28 kg / m²
* Blood typing identical to the recipient
* Absence of significant medical, psychiatric problems or previous abdominal surgery
* Normal laboratory tests: liver function tests, blood count, coagulogram, pregnancy test and serology for hepatitis B, C and HIV
* Normal imaging exams: CT of the abdomen and pelvis with liver volume (remaining volume - 30-40% of the total liver volume), MRI with cholangioresonance

Exclusion Criteria:

* ERCP candidates (case group)

  * Use of antibiotics during ERCP or in the last 2 months prior to the procedure
  * Emergency ERCP
  * Pregnancy
  * Uncorrected coagulopathy

Liver transplant living-donor (control group)

* Use of antibiotics in the last 2 months prior to the procedure
* Pregnancy
* Uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary care adult patients with hepatobiliopancreatic diseases compared to healthy people, that are living donors of liver transplant
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-16 (Estimated)

PRIMARY OUTCOMES:
Composition of the biliary microbiota | 2 years
  In this study, the investigator's objective will be to characterize the specific composition of the biliary microbiota in patients with hepatobiliopancreatic diseases in comparison with healthy people using 16S ribosomal RNA (rRNA) pyrosequencing methods.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo School of Medicine, São Paulo, Brazil

REFERENCES:
- [Derived] Nascimento FSD, Suzuki MO, Taba JV, de Mattos VC, Pipek LZ, D'Albuquerque EMC, Iuamoto L, Meyer A, Andraus W, Pinho JRR, de Moura EGH, Setubal JC, Carneiro-D'Albuquerque LA. Analysis of biliary MICRObiota in hepatoBILIOpancreatic diseases compared to healthy people [MICROBILIO]: Study protocol. PLoS One. 2020 Nov 19;15(11):e0242553. doi: 10.1371/journal.pone.0242553. eCollection 2020. PMID 33211762

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT04391426/Prot_002.pdf
  • Informed Consent Form (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT04391426/ICF_001.pdf